CLINICAL TRIAL: NCT03506971
Title: Evaluate the Effects of a Preventive Care at Home on Young Child's Development
Brief Title: Early Childhood : Action Research in the Lunévillois Area (PERL)
Acronym: PERL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: Conseil Départemental, Protection Maternelle Infantile :PMI, France (Unknown); Agence Regionale de Sante d'Ile de France (Other Government); Family Allowance Fund, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIPH 2017-01; IDRCB 2017-A00896-47 (Other: ANSM (French competent authority))
Record Dates: First submitted 2018-02-16; First posted 2018-04-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Development, Infant; Perinatal Disorder
Keywords: Young child's development; Home visits; Early interactions; attachment; parenthood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants (Experimental): As part of this research, families will benefit from
  * "pediatric nurse's interventions" : home visits by a pediatric nurse who will center around three times: a time of observation of the development and progress of the baby, a time for play with the baby and a time to listening the parents.
  * "psychologist's evaluation" and "joint home visits" : home visits by the coordinating psychologist to evaluate three areas: child development, parenthood and parent-child interaction.
  Interventions: Other: Pediatric Nurse's interventions; Other: Joint home visits
- Control (Other): "psychologist's evaluation" : home visits by the coordinating psychologist to evaluate three areas: child development, parenthood and parent-child interaction.
  Interventions: Other: Psychologist's evaluation

INTERVENTIONS:
Other: Psychologist's evaluation — The research coordinator psychologist will evaluate: the development of the baby, the early interactions between the baby and his mother, attachment, maternal psychiatric symptoms, the experience of parenting and maternal sensitivity.
  Arms: Control
Other: Pediatric Nurse's interventions — Pediatrics nurses perform preventive home visits that are based on : joint observation with the parents of the baby, play with the baby and his parents, interview with the parents on their parenthood
  Rhythm of home visits:
  * 1 every month from birth to 1 year
  * 1 every 2 months from 1 year to 2 years
  * 1 every 3 months from 2 years to 4 years
  Arms: Participants
Other: Joint home visits — Coordinating psychologist and the referent pediatric nurse will perform home visits. During this time, the psychologist evaluate : the development of the baby, the early interactions between the baby and his mother, attachment, maternal psychiatric symptoms, the experience of parenting and maternal sensitivity.
  Rhythm of joint home visits:
  * 1 at 4 months
  * 1 at 24 months
  Arms: Participants

SUMMARY:
The PERL project is a research in prevention in perinatality. The objective of this research is to offer preventive and regular care at familie's home in the Lunévillois area, while integrating it into the existing practices of the maternal and child protection, in the framework of a partnership between the PMI (Protection Maternal Infantile) and the child psychiatry.

An innovative prevention device to support the interactions and development of the child will be proposed to about sixty families, randomly recruited into the general population.

If the family agrees to participate, their will benefit from regular home visits by a pediatric nurse, accompanied on certain times by a psychologist, for a period of 4 years from the birth of the child.

This home-visits accompaniment, centered on listening and observation, focuses on three areas: baby's development, parenthood and parent-child's interactions.

A longitudinal and comparative evaluation will be carried out with a "control" group recruited according to the same conditions and at the same time as the "participants" group.

A parallel research on the processes and mechanism will be carried out in partnership with the School of Public Health in order to define and validate the intervention theory (what are the mobilized levers produced and how, what are the mechanisms linking the intervention to its results), to describe the implementation and the processes involved, and to analyze the effects of context, especially social, on processes and results.

ELIGIBILITY:
Inclusion Criteria:

* Parents living in the Lunevillois area
* Mother to be 8 months pregnant
* Baby who's born from january to december 2018

Exclusion Criteria:

* No exclusion criteria

Ages: 1 Minute to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Brunet-Lézine-revised test : assessment of change between 3 and 24 months and between two groups of the study. | 3 and 24 months
  Assessment of children psychomotor development. This test can be used at any time from the age of 0 to 30 months
ADBB (Alarm Distress BaBy) : assessment of change between 3 and 24 months and between two groups of the study. | 3 and 24 months
  Filmed evaluation of relational withdrawal of young children. This evaluation can be used at any time from the age of 2 to 24 months
EPDS : Edinburgh Postnatal Depression Scale | 3 months
  The Edinburgh Postnatal Depression Scale (EPDS) is a set of 10 screening questions that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child.
  To complete this set of questions, the parent should select the number next to the response that comes closest to how they have felt in the past seven days.
  The total score is calculated by adding the numbers selected for each of the 10 items. If the parent's score is 10 points or above, they should speak to a health professional about those symptoms.
ERP (Entretien sur les représentations Parentales, no traduction for acronym): assessment of change between 3 and 24 months and between two groups of the study. | 3 and 24 months
  Interview on Parent's Representations
ERTL 4 : Epreuve de repérage des Troubles du Langage = French questionnaire. No traduction for acronym | 4 YEARS
  Test of Spotting of language delays at 4 years, carried out in a systematic way by the teams of maternal and child protection
Q-SORT attachment | 24 months
  Q-SORT for evaluate the attachment
Mini-MBQS (Maternal Behavior Q-Sort ) : assessment of change between 3 and 24 months and between two groups of the study. | 3 and 24 Months
  25 items to obtain an assessment of global maternal sensitivity
BDI : Beck Depression Inventory (13 items) | 24 Months
  This is a multiple-choice self-report inventory for measuring the severity of depression
SCL-90R (Symptom Checklist-90-R) : assessment of change between 3 and 24 months and between two groups of the study. | 3 and 24 Months
  Symptom check-list, self-assessment questionnaire for psychiatric symptoms
BITSEA : Brief Infant Toddler Social and Emotional Assessment | 24 months
  Early screening of social and emotional difficulties or developmental delays for children. This assessment can be used at any time from the age of 12 to 36 months.
HAQ : Helping Alliance Questionnaire | 3 months
  Evaluate the therapeutic alliance
HAQ | 24 months
  Helping Alliance Questionnaire, to evaluate the therapeutic alliance
Bobigny's early childhood interactions assessment | 3 months
  It's an assessment of early childhood interactions baby-mother
Bobigny's early childhood interactions assessment | 24 months
  It's an assessment of early childhood interactions baby-mother

SECONDARY OUTCOMES:
FAS : Family Affluence Scale | 3 and 24 Months
  Small questionnaire to describe family's affluence. 4 questions asked : How many computers do you have at home ? (none, 1, 2, more than 2) / Do you have a car at home? (no, 1, 2 or more) / Do you have your own bedroom at home? (yes, no) / For the last 12 months, how many times have you travelled with your family for holidays? (never, once, twice, more than twice) Assessment of change will be done between 3 and 24 months and between two groups of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BUCHHEIT, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchheit S, Kabuth B, Colombo MC, Ligier F. Child Development and Early Interaction: PERL Research Protocol, a Preventive Home Visiting Program, Randomized Controlled Trial in France. Front Psychiatry. 2021 Jun 30;12:641468. doi: 10.3389/fpsyt.2021.641468. eCollection 2021. PMID 34276432